CLINICAL TRIAL: NCT06867237
Title: The Effect of Continuous Management of Suction Cuff Pressure and Subglottic Irrigation Suction on the Outcomes of Mechanically Ventilated Patients With High Risk of Aspiration: a Single-center, Prospective, Randomized Controlled Trial
Brief Title: The Effect of Continuous Management of Suction Cuff Pressure and Subglottic Irrigation Suction on Preventing VALRI Study
Acronym: SCOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, Doctor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2025-070
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Ventilation Acquired Pneumonia
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suction cuff pressure and suction intervention (Active Comparator)
  Interventions: Device: Suction cuff pressure
- Standard care (No Intervention)

INTERVENTIONS:
Device: Suction cuff pressure — Use the device to do continuous management of suction cuff pressure and subglottic irrigation suction
  Other Names: airway management
  Arms: Suction cuff pressure and suction intervention

SUMMARY:
Assessing the effectiveness of continuous cuff pressure management combined with subglottic suction irrigation in reducing ventilator-associated lower respiratory tract infections (VALRTI) in mechanically ventilated patients at high risk of aspiration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Undergoing endotracheal intubation or tracheostomy;
3. Expected duration of mechanical ventilation exceeding 72 hours;
4. Presence of one or more high-risk factors for reflux/aspiration: recurrent laryngeal nerve injury, cerebral infarction/cerebral hemorrhage (new or pre-existing swallowing dysfunction), cranial surgery/traumatic brain injury (TBI), neuromuscular junction disorders (e.g., myasthenia gravis, muscular dystrophy, Parkinson's disease, or other conditions that weaken swallowing muscle strength and coordination), continuous use of muscle relaxants for ≥ 48 hours during mechanical ventilation, ICU-acquired myopathy, ICU-acquired weakness, gastroparesis (gastric residual volume > 500 mL/6 hours), or impaired consciousness;
5. Voluntary participation in the study by the subject or their legal representative, with signed informed consent.

Exclusion Criteria:

1. Expected duration of mechanical ventilation less than 48 hours;
2. Pregnant or breastfeeding women;
3. Patients with tracheoesophageal or bronchopleural fistula;
4. Difficult intubation (more than three attempts) or patients with reflux/aspiration during intubation (with lung injury and secondary pulmonary infection);
5. Patients with irreversible disease, end-stage conditions, or those expected to die in the near future;
6. Patients already diagnosed with ventilator-associated pneumonia (VAP), i.e., excluding hospital-acquired pneumonia;
7. Patients participating in other clinical trials that are expected to influence the results of this study;
8. Patients deemed unsuitable for inclusion in the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of days free from VALRTI within 28 days. | 28 days
  The number of days free from ventilator-associated lower respiratory tract infection (VALRTI) within 28 days.

IPD SHARING:
Plan to Share IPD: Undecided